CLINICAL TRIAL: NCT05429177
Title: This is a Phase I, Randomized, Double-blind, Vehicle-controlled Study of QY101 Ointment in Chinese Healthy Subjects
Brief Title: A First-in-Human Study of QY101 Ointment in Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: E-nitiate Biopharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QY101-Ⅰ-1
Record Dates: First submitted 2022-06-08; First posted 2022-06-23 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- SAD Cohort 1(0.1% QY101 ointment or vehicle apply to 5%BSA) (Experimental): 3 subjects use 0.1% QY101 ointment，1 subject uses vehicle topical applied to 5% Body Surface Area，assessed until 72 hours postdose
  Interventions: Drug: QY101 ointment or vehicle
- SAD Cohort 2(0.1% QY101 ointment or vehicle apply to 20%BSA) (Experimental): 6 subjects use 0.1% QY101 ointment，2 subjects use vehicle topical applied to 20% Body Surface Area，assessed until 72 hours postdose
  Interventions: Drug: QY101 ointment or vehicle
- SAD Cohort 3(0.3% QY101 ointment or vehicle apply to 20%BSA) (Experimental): 6 subjects use 0.3% QY101 ointment，2 subjects use vehicle topical applied to 20% Body Surface Area，assessed until 72 hours postdose
  Interventions: Drug: QY101 ointment or vehicle
- SAD Cohort 4(0.5% QY101 ointment or vehicle apply to 20%BSA) (Experimental): 6 subjects use 0.5% QY101 ointment，2 subjects use vehicle topical applied to 20% Body Surface Area，assessed until 72 hours postdose
  Interventions: Drug: QY101 ointment or vehicle
- SAD Cohort 5(1.0% QY101 ointment or vehicle apply to 20%BSA) (Experimental): 6 subjects use 1.0% QY101 ointment，2 subjects use vehicle topical applied to 20% Body Surface Area，assessed until 72 hours postdose
  Interventions: Drug: QY101 ointment or vehicle
- SAD Cohort 6(1.0% QY101 ointment or vehicle apply to 40%BSA) (Experimental): 6 subjects use 1.0% QY101 ointment，2 subjects use vehicle topical applied to 40% Body Surface Area，assessed until 72 hours postdose
  Interventions: Drug: QY101 ointment or vehicle
- MAD Cohort 7(0.3% QY101 ointment or vehicle apply to 20%BSA) (Experimental): 6 subjects use 0.3% QY101 ointment，2 subjects use vehicle topical applied to 20% Body Surface Area，twice daily for 7 days and once in the morning on D8
  Interventions: Drug: QY101 ointment or vehicle
- MAD Cohort 8(0.5% QY101 ointment or vehicle apply to 20%BSA) (Experimental): 6 subjects use 0.5% QY101 ointment，2 subjects use vehicle topical applied to 20% Body Surface Area，twice daily for 7 days and once in the morning on D8
  Interventions: Drug: QY101 ointment or vehicle
- MAD Cohort 9(1.0% QY101 ointment or vehicle apply to 20%BSA) (Experimental): 6 subjects use 1.0% QY101 ointment，2 subjects use vehicle topical applied to 20% Body Surface Area，twice daily for 7 days and once in the morning on D8
  Interventions: Drug: QY101 ointment or vehicle
- MAD Cohort 10(1.0% QY101 ointment or vehicle apply to 40%BSA) (Experimental): 6 subjects use 1.0% QY101 ointment，2 subjects use vehicle topical applied to 40% Body Surface Area，twice daily for 7 days and once in the morning on D8
  Interventions: Drug: QY101 ointment or vehicle

INTERVENTIONS:
Drug: QY101 ointment or vehicle — QY101 ointment or vehicl topical applied to skin

SUMMARY:
This is a phase I, randomized, double-blind, vehicle-controlled，single and multiple ascending dose study to assess the safety, tolerability, and pharmacokinetics of QY101 ointment in Chinese healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. The subjects were fully aware of the purpose, nature, methods and possible adverse reactions of the trial, volunteered as subjects, and signed an informed consent form before the start of any research process.
2. Male and female subjects aged 18 to 45 (including 18 and 45).
3. Male weight≥50.0 kg, female weight≥45.0 kg; BMI is in the range of 19.0 ~ 26.0 kg/ m2 (including the critical value).
4. The subjects had no history of chronic or serious diseases such as cardiovascular, liver, kidney, respiration, blood and lymph, endocrine, immune, mental, nervous, gastrointestinal system, and were in good health.
5. Physical examination, vital signs, clinical laboratory examination values (blood routine, urine routine, blood biochemistry, blood coagulation function, stool routine and occult blood, pregnancy test (female), hepatitis, HIV, syphilis), 12-lead ECG, chest X-ray examination, abdominal ultrasound examination results are all within the normal range or abnormalities with no clinical significance.
6. The subjects (including male subjects) had no fertility plan, voluntary use of effective contraception and no plan to donate sperm or eggs during the screening period and within 6 months after the end of the last administration.
7. The subjects were able to communicate well with the researchers and understand and comply with the requirements of this study.

Exclusion Criteria:

1. Allergic constitution, such as a history of allergy to two or more drugs and food, or those known to be allergic to QY101 and excipients.
2. Screen those who have undergone surgery within the previous 3 months, or who plan to undergo surgery during the study period, or who have undergone surgery that will affect the absorption, distribution, metabolism and excretion of drugs.
3. Diseases that need to be excluded with abnormal clinical manifestations, including, but not limited to, diseases of the nervous system, cardiovascular system, blood and lymphoid system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolic and skeletal system, etc.
4. Subjects who cannot tolerate venipuncture, have a history of dizzy needles and blood sickness.
5. Subjects with a history of severe skin disease (subject to the judgment of the researcher).
6. Live (attenuated) vaccine was vaccinated within 2 months before screening.
7. Smoking or drinking within 3 months before screening (smoking: > 10 cigarettes per day; drinking: > 15g pure alcohol per day, equivalent to 450mL beer, 150mL wine or 50mL low alcohol), or positive for nicotine, alcohol, abuse drugs (morphine / methamphetamine / ketamine / dimethylene dioxyamphetamine / tetrahydrocannabinic acid).
8. Screen subjects who have participated in other drug clinical trials or have not come to participate in clinical trials within the first 3 months.
9. Non-physiological blood loss ≥ 200ml within 3 months before screening (including trauma, blood collection, blood donation), or plan to donate blood during the study period or within 1 month after the end of the study.
10. The subjects (female) are lactating.
11. Strong inhibitors or inducers of CYP3A liver metabolic enzymes were used in the previous 2 weeks (see Appendix 2 for details), or any drugs, including prescription, over-the-counter and herbal medicines, were used for oral or topical use, except vitamins and / or paracetamol.
12. To screen subjects who drank too much tea, coffee and / or caffeinated beverages (more than 8 cups, 1 cup = 250mL) every day for the first 3 months.
13. Subjects with abnormal vital signs were included in the standard reference range (including critical value): sitting systolic blood pressure 90~139mmHg, diastolic blood pressure 55-89mmHg, pulse 55-100bpm, body temperature 36.037.4C, breathing 12-22bpm; if the subject's first examination result is abnormal, retest can be carried out after rest.
14. There are tattoos, birthmarks, sunburns, abrasions, ulcers, erythema, dryness, scabs and scars in the target area (back, abdomen and lower limbs from thigh to calf) of the subjects.
15. Subjects determined by other researchers to be unfit to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | SAD：Day1 to Day18；MAD：Day1 to Day25
Number of Participants With Clinical Laboratory Abnormalities | SAD：Screening period and Day4；MAD：Screening period, Day5 and Day11
Number of Participants With Clinically Significant Changes Form Baseline in Vital Signs | SAD：Screening period and Day1 to Day4；MAD：Screening period and Day1 to Day11
Severity of local skin irritation | SAD：Day1 to Day4；MAD：Day1 to Day11
  Skin irritation response assessment recording method: -: no reaction; + (mild): only erythema can be observed; + (moderate): moderate erythema, edema; + (severe): severe erythema, edema with papules, vesicles; + (severe): severe erythema, edema, bullae, and even necrosis.
Number of Participants With Clinically Significant Treatment-emergent Electrocardiogram (ECG) Findings | SAD：Screening period and Day4；MAD：Screening period, Day5 and Day11
Number of Participants With Clinically Significant Changes Form Baseline in Physical Examination | SAD：Screening period and Day4；MAD：Screening period, Day5 and Day11

SECONDARY OUTCOMES:
Tmax of QY101 | SAD：Day1 to Day4；MAD：Day1，Day5 to Day11
  Time of maximum concentration
Cmax of QY101 | SAD：Day1 to Day4；MAD：Day1，Day5 to Day11
  Maximum observed plasma concentration
t1/2 of QY101 | SAD：Day1 to Day4；MAD：Day1，Day5 to Day11
  The time it takes for the blood concentration of the drug to drop by half from the highest value in the body
AUC0-∞ of QY101 | SAD：Day1 to Day4；MAD：Day1，Day5 to Day11
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration

CONTACTS AND LOCATIONS:
Overall Officials: zourong ruan, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No